CLINICAL TRIAL: NCT06566495
Title: Reusable Tourniquets as Potential Risk of Microbial Transmission - Comparison of Operating Theatre and Emergency Department
Brief Title: Microorganisms on Reusable Tourniquets
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: KB/45/2024
Record Dates: First submitted 2024-08-14; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Microbial Colonization; Infection, Bacterial; HAI; Nurse's Role; Vascular Access Device Complications; Vascular Access Complication; CRBSI - Catheter Related Bloodstream Infection; Catheter Infection; Device Colonisation
Keywords: Tourniquet; Cross Infection; Vascular Access Devices; Infection Control
MeSH Terms: conditions — Communicable Diseases; Bacterial Infections; Cross Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- reusable tourniquets used by indefinite time: 6 tourniquets from emergency department and 11 tourniquets from operating theatre
  Interventions: Device: collection of microbiological material from reusable tourniquets
- reusable tourniquets used by 14 days: 6 tourniquets from emergency department and 14 tourniquets from operating theatre
  Interventions: Device: collection of microbiological material from reusable tourniquets
- reusable tourniquets used by 28 days: 6 tourniquets from emergency department and 10 tourniquets from operating theatre
  Interventions: Device: collection of microbiological material from reusable tourniquets

INTERVENTIONS:
Device: collection of microbiological material from reusable tourniquets — Microbiological analysis
  The material was collected in each group in the same way.
  Other Names: sampling of microbiological material

SUMMARY:
The purpose of this study was to compare microbial contamination on the surface of reusable stasis after indefinite use, 2 weeks and 4 weeks. We investigated how the site - the operating theater and the emergency department, as well as the time of use - affects the number of organisms.

DETAILED DESCRIPTION:
The cross-sectional study was conducted in the operating theater and emergency department of a tertiary referral hospital in Gdansk, Poland, in three part from March to April 2024. The study included reusable tourniquets used by the hospital's medical staff during vascular access generation.

After each stage of the in-hospital study, the stasis was collected and replaced with new ones. A total of 53 reusable stasis were collected in three phases of the study and were subjected to microbiological analysis at the Department of Immunobiology and Environmental Microbiology of the Medical University of Gdansk. The tourniquets were collected into disposable, sterile bags. In the first stage of the study, tourniquets were collected of indefinite use (n= 17). In the second and third stages of the study, stasis used for 14 (n=20) and 28 (n=16) days, respectively, were collected. All tourniquets were labeled and assigned to different rooms located within the surveyed wards. The trial was conducted separately, for the plastic fastener and the fabric band. The plastic parts of the tourniquets were placed in sterile glass dishes. Under laboratory conditions, the plastic parts of the stasis were cut off and placed in the dishes. Using sterile swabs soaked in 0.9% sodium chloride, the plastic was swabbed, after which the tip of the swab was cut off, placed in a tube with 0.9% sodium chloride (3ml), which was shaken in a Vortex device (30 seconds) and the obtained material was seeded on columbia Agar with 5% sheep blood. The material part of the stasis was placed in a sterile homogenization bag with the addition of 100ml of nutrient broth. The bag was then placed in a Stomacher Homogenizer for two minutes to detach the microorganisms from the porous surface of the material. The resulting homogenate was transferred in a concentrated state and diluted tenfold using 200 μl pipettes onto columbia Agar media supplemented with 5% sheep blood.200 μl of concentrated homogenate was seeded onto the quality growth media MacConkey Broth, King B Agar, CHROMagar E. coli and other coliforms. The protected material was incubated for 24 hours at 37°C, in an aerobic atmosphere. After this time, bacterial colonies were counted and counts were performed to determine the number of microorganisms on the surface of the stasis (CFU/cm2). Due to the assumptions of the experiment and the time frame, eight tourniquets were not included in the analysis. From the information obtained from the medical staff, this was due to significant soiling, making it impossible to use the tourniquets, and in a few cases the plastic fastener broke.

ELIGIBILITY:
Inclusion Criteria:

* reusable tourniquets used to make the vessel visible

Exclusion Criteria:

* disposable tourniquets used to make the vessel visible

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 53 reusable tourniquets
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Standard Deviation and median of colony forming units (CFU/cm2) in the emergency department | 24 hours
  After 24h incubation at 37 deg C, we evaluated the number of bacterial colony-forming colonies on leaf and quality plates. The average number of CFU/cm2 in all stages of the study for the emergency department is 19,110, 34 CFU/cm2. For the MCC substrate for the emergency department medium 227.65; standard deviation 102.75 CFU/cm2. For the King B substrate for the emergency department medium 241.71, standard deviation 115.15 18 CFU/cm2. There is no statistically significant difference for OD versus CFU/cm2 during the second and third intake. There were no bacterial growth was obtained on the ECC plate.
Standard Deviation and median of colony forming units (CFU/cm2) in the operating theatre | 24 hours
  After 24h incubation at 37 deg C, we evaluated the number of bacterial colony-forming colonies on leaf and quality plates. The average number of CFU/cm2 in all stages of the study for the operating theatre was 88.27 CFU/cm2. For the MCC substrate for the operating theatre medium 14.18 standard deviation 24.06 CFU/cm2. For the King B substrate for the operating theatre medium 33.07 standard deviation 65.18 CFU/cm2.There is no statistically significant difference for OD versus CFU/cm2 during the second and third intake. There were no bacterial growth was obtained on the ECC plate.

SECONDARY OUTCOMES:
Blood stains and CFU | 2 months
  23 of 53 examined tourniquets (43%), 12/18 (67%) from the emergency department and 11/35 (31%) from the operating theatre had visible blood stains. Blood stains did not affect the number of colony-forming units (CFUs).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Univeristy of Gdańsk, Gdansk, Dębinki Street, Poland